CLINICAL TRIAL: NCT06690567
Title: Clinical Outcomes of Contemporary IMPELLA Devices in Cardiogenic Shock and High-risk Percutaneous Coronary Intervention
Acronym: IMMERGE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, Medical Doctor, University of Turin, Italy
Other Study IDs: IMMMERGE
Record Dates: First submitted 2024-11-04; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2023-12

CONDITIONS: Cardiogenic Shock; PCI Patients; Mechanical Circulatory Support
Keywords: IMPELLA; CARDIOGENIC SHOCK; COMPLEX PCI
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with cardiogenic shock or patients undergoing complex PCI, with Impella implantation: Impella implantation as only intervention needed
  Interventions: Device: Impella implantation

INTERVENTIONS:
Device: Impella implantation — To implante Impella

SUMMARY:
The IMMERGE registry is an observational, international multicentric study, including patients underwent IMPELLA implantation in the participating centers both for cardiogenic shock and high-risk PCI. Only IMPELLA CP, 5.0 and 5.5 devices will be included. Consecutive patients with CS and CHIPs implanted with Impella® CP, 5.0 and 5.5 with at least 6 months of follow-up completed will be enrolled in the registry. Baseline clinical and echocardiographic variables, peri-procedural haemodynamic parameters, laboratoristic findings and complications, together with follow-up outcomes data will be recorded in a dedicated database.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 18 years-old with CS or CHIPs
* Impella® device implanted (CP, 5, 5.5)

Exclusion Criteria:

* Age < 18 years
* No Impella implanted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paitents with cardiogenic shock or CHIP-PCI who underwent Impella device implantation
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
long-term overall mortality | 12 months

SECONDARY OUTCOMES:
30-day overall and cardiovascular mortality | 30 day
Rate of acute kidney injury (AKIN classification) and need for renal replacement therapy (RRT) | 12 months
Rate of bleedings according to the BARC classification | 12 months
Rate of vascular complications, limb-ischemia, hemolysis (INTERMACS definition) | 12 months
Rate of neurological events (stroke and TIA) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy, Italy

REFERENCES:
- [Background] O'Neill WW, Anderson M, Burkhoff D, Grines CL, Kapur NK, Lansky AJ, Mannino S, McCabe JM, Alaswad K, Daggubati R, Wohns D, Meraj PM, Pinto DS, Popma JJ, Moses JW, Schreiber TL, Magnus Ohman E. Improved outcomes in patients with severely depressed LVEF undergoing percutaneous coronary intervention with contemporary practices. Am Heart J. 2022 Jun;248:139-149. doi: 10.1016/j.ahj.2022.02.006. Epub 2022 Feb 19. PMID 35192839
- [Background] O'Neill WW, Kleiman NS, Moses J, Henriques JP, Dixon S, Massaro J, Palacios I, Maini B, Mulukutla S, Dzavik V, Popma J, Douglas PS, Ohman M. A prospective, randomized clinical trial of hemodynamic support with Impella 2.5 versus intra-aortic balloon pump in patients undergoing high-risk percutaneous coronary intervention: the PROTECT II study. Circulation. 2012 Oct 2;126(14):1717-27. doi: 10.1161/CIRCULATIONAHA.112.098194. Epub 2012 Aug 30. PMID 22935569
- [Background] Chieffo A, Ancona MB, Burzotta F, Pazzanese V, Briguori C, Trani C, Piva T, De Marco F, Di Biasi M, Pagnotta P, Casu G, Giustino G, Montorfano M, Pappalardo F, Tarantini G; Collaborators. Observational multicentre registry of patients treated with IMPella mechanical circulatory support device in ITaly: the IMP-IT registry. EuroIntervention. 2020 Feb 7;15(15):e1343-e1350. doi: 10.4244/EIJ-D-19-00428. PMID 31422925
- [Background] Dhruva SS, Ross JS, Mortazavi BJ, Hurley NC, Krumholz HM, Curtis JP, Berkowitz A, Masoudi FA, Messenger JC, Parzynski CS, Ngufor C, Girotra S, Amin AP, Shah ND, Desai NR. Association of Use of an Intravascular Microaxial Left Ventricular Assist Device vs Intra-aortic Balloon Pump With In-Hospital Mortality and Major Bleeding Among Patients With Acute Myocardial Infarction Complicated by Cardiogenic Shock. JAMA. 2020 Feb 25;323(8):734-745. doi: 10.1001/jama.2020.0254. PMID 32040163
- [Background] Schrage B, Ibrahim K, Loehn T, Werner N, Sinning JM, Pappalardo F, Pieri M, Skurk C, Lauten A, Landmesser U, Westenfeld R, Horn P, Pauschinger M, Eckner D, Twerenbold R, Nordbeck P, Salinger T, Abel P, Empen K, Busch MC, Felix SB, Sieweke JT, Moller JE, Pareek N, Hill J, MacCarthy P, Bergmann MW, Henriques JPS, Mobius-Winkler S, Schulze PC, Ouarrak T, Zeymer U, Schneider S, Blankenberg S, Thiele H, Schafer A, Westermann D. Impella Support for Acute Myocardial Infarction Complicated by Cardiogenic Shock. Circulation. 2019 Mar 5;139(10):1249-1258. doi: 10.1161/CIRCULATIONAHA.118.036614. PMID 30586755
- [Background] Geller BJ, Sinha SS, Kapur NK, Bakitas M, Balsam LB, Chikwe J, Klein DG, Kochar A, Masri SC, Sims DB, Wong GC, Katz JN, van Diepen S; American Heart Association Acute Cardiac Care and General Cardiology Committee of the Council on Clinical Cardiology; Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Peripheral Vascular Disease; and Council on Cardiovascular Surgery and Anesthesia. Escalating and De-escalating Temporary Mechanical Circulatory Support in Cardiogenic Shock: A Scientific Statement From the American Heart Association. Circulation. 2022 Aug 9;146(6):e50-e68. doi: 10.1161/CIR.0000000000001076. Epub 2022 Jul 7. PMID 35862152
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- [Background] Potapov EV, Antonides C, Crespo-Leiro MG, Combes A, Farber G, Hannan MM, Kukucka M, de Jonge N, Loforte A, Lund LH, Mohacsi P, Morshuis M, Netuka I, Ozbaran M, Pappalardo F, Scandroglio AM, Schweiger M, Tsui S, Zimpfer D, Gustafsson F. 2019 EACTS Expert Consensus on long-term mechanical circulatory support. Eur J Cardiothorac Surg. 2019 Aug 1;56(2):230-270. doi: 10.1093/ejcts/ezz098. PMID 31100109
- [Background] Lauten A, Engstrom AE, Jung C, Empen K, Erne P, Cook S, Windecker S, Bergmann MW, Klingenberg R, Luscher TF, Haude M, Rulands D, Butter C, Ullman B, Hellgren L, Modena MG, Pedrazzini G, Henriques JP, Figulla HR, Ferrari M. Percutaneous left-ventricular support with the Impella-2.5-assist device in acute cardiogenic shock: results of the Impella-EUROSHOCK-registry. Circ Heart Fail. 2013 Jan;6(1):23-30. doi: 10.1161/CIRCHEARTFAILURE.112.967224. Epub 2012 Dec 4. PMID 23212552